CLINICAL TRIAL: NCT00881283
Title: Role of Adipokines in Long-term Cardiovascular Risk in Cured Cushing's Patients
Brief Title: Long-term Cardiovascular Risk in Cured Cushing's Patients
Status: Terminated | Type: Observational
Why Stopped: Decision made to close study early.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Other Study IDs: 2008-p-001379
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Cushing's Disease
Keywords: Cushing's disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cured Cushing's disease

SUMMARY:
The purpose of this study is to determine whether subjects who have been affected by Cushing's disease in the past maintain some different characteristics compared with subjects who have never been diagnosed with the disease.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been cured of Cushing's disease at least 5 years ago.

Exclusion Criteria:

* patients who have been cured of Cushing's disease more than 15 years ago.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cured Cushing's disease
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-09-08 (Actual); Primary Completion 2010-03-30 (Actual); Study Completion 2010-03-30 (Actual)

PRIMARY OUTCOMES:
adipokine measurements | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Neuroendocrine Clinical Center, Boston, Massachusetts, United States